CLINICAL TRIAL: NCT00064519
Title: Genetics of CRP in Families With Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ulrich Broeckel MD, Professor of Pediatrics, Medical College of Wisconsin
Other Study IDs: 1225; R01HL074321 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-10 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — i.) Blood: A blood sample (30 cc, ~2 tablespoons) will be drawn. This will take place in the catheterization lab at the end of the catheterization procedure or by using standard venipuncture technique during a clinic visit or at community outreach events when feasible.
  ii.) Buccal Swab: The participant uses specially prepared cotton swabs (called buccal swabs) to rub in a circular motion on the inside of both cheeks. The swabs collect cheek cells that can be processed to obtain DNA.
  iii.) Saliva: A saliva sample is obtained by having the participant spit in a special vial specifically designed for genetic testing. The participant will continue to spit into the vial until it contains 2 ml (about 1 teaspoon) of saliva.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Families with MI: In conjunction with collaborators in Germany, we have established one of the largest collections of families with MI, comprising 1,406 individuals in 513 Western-European families. Based on this collection, our total genome scan and linkage analysis has identified a region on chromosome 14 with a significant linkage signal for myocardial infarction (LOD = 3.9, pointwise P = 0.00015, genome-wide P < 0.05)5. Preliminary results from an association study in a subset of these families has identified a small set of single nucleotide polymorphisms (SNPs) within candidate genes in this region as being suggestively associated with MI.
  No drugs are to be administre

SUMMARY:
To investigate the genetics of C reactive protein in families with myocardial infarction.

DETAILED DESCRIPTION:
BACKGROUND:

Coronary artery disease (CAD) and myocardial infarction (MI) are the leading causes of death in the Western world. Numerous epidemiological studies have demonstrated the impact of various risk factors, such as arterial hypertension, hypercholesterolemia and diabetes mellitus. While these risk factors are partly under genetic control, a positive family history remains an additional independent predictor of CAD, suggesting the presence of as yet unidentified susceptibility loci. Given the enormous public health burden of CAD, there is significant interest in identifying its specific genetic foundations. As intensive experimental investigations continue, the inflammatory component of the disease process leading to atherosclerosis evolves as a key aspect in the disease process. Recent evidence demonstrates that systemic markers of inflammation such as C reactive protein (CRP) can predict those at high risk of coronary events. CRP emerges with much attention as both a diagnostic marker and therapeutic target with serum levels determined to a significant extent by genetic factors.

DESIGN NARRATIVE:

To elucidate the genetic basis of the inflammatory component of myocardial infarction and the regulation of C reactive protein, a gene function oriented evaluation of candidate genes will be conducted. Therefore the specific aims are as follows, 1. Identify positional candidate genes within regions identified for MI and CRP which are functionally related to inflammation and inflammatory processes. Sequence variation in selected candidate genes will be identified. 2. Evaluate the effect of these variants with regard to MI and CRP in two different ethnic populations: a family set of European Caucasians and a population-based, Hispanic family dataset. The role of CRP will be evaluated as a predictor of cardiovascular events in the study populations. Since clinical follow up data are available on both study populations, the extent to which CRP contributes to an increased risk for cardiovascular events will be analyzed.

ELIGIBILITY:
1. First Part DNA Collection

   a.) Inclusion Criteria i.) Being 18 years of age or older. ii.) Having had a cardiac catheterization procedure performed or undergoing one in the near future.

   iii.) A person having a family history of coronary artery disease and having at least one family member that has had a cardiac catheterization that is willing to participate.

   iv.) Having coronary artery (right, left main, circumflex, marginal and/or diagonal) blockage in a specific portion of the vessel (ostial, proximal, mid and/or distal).

   b.) Exclusion Criteria i.) Having had a bone marrow transplant.
2. Second Part Coronary Collateralization and Extended Phenotyping a.) Inclusion Criteria i.) Having participated in DNA collection. ii.) Having at least one coronary artery with 100% blockage or iii.) Having normal coronary arteries with no blockage b.) Exclusion Criteria i.) Having received a diagnosis and treatment for kidney disease, cancer, myocardial infarction within the last three (3) months.

ii.) Having a heart transplant.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals having CAD and individuals not having CAD
Sampling Method: Non-Probability Sample
Enrollment: 1406 (Actual)
Dates: Start 2003-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Association of markers with cardiovascular event | Event recorded at time of recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Broeckel, Principal Investigator — Medical College of Wisconsin